CLINICAL TRIAL: NCT02062346
Title: The Vascular Effects of Endothelin Receptor Antagonism in Systemic Vasculitis
Brief Title: Endothelin Antagonism in ANCA Vasculitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Bean ICRF clinical study
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Vasculitis
Keywords: endothelin;; blood pressure;; vasculitis
MeSH Terms: conditions — Vasculitis | interventions — cyclo(Trp-Asp-Pro-Val-Leu); Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Saline placebo
  Interventions: Drug: Placebo
- BQ123 (Experimental): Intravenous infusion of BQ123 1000nmol/min for 15min
  Interventions: Drug: BQ123
- BQ123/788 (Experimental): Intravenous infusion of BQ123 1000nmol/min and BQ788 300nmol/min
  Interventions: Drug: BQ123/788
- Assessment of forearm vascular function (No Intervention): Response of forearm blood flow to endothelium-dependent and endothelium-independent vasodilators

INTERVENTIONS:
Drug: BQ123 — Intravenous infusion of BQ123 ( selective ETA antagonist )
  Other Names: Selective ETA antagonism
  Arms: BQ123
Drug: BQ123/788 — or BQ123/788 (mixed ETA/B antagonists)
  Other Names: mixed ETA/B antagonism
  Arms: BQ123/788
Drug: Placebo — Intravenous infusion of saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Patients with vasculitis commonly develop cardiovascular disease. The reasons for this are not clear and is not adequately treated with current drugs. It is thus understand the reasons why patients with vasculitis develop cardiovascular disease in order to develop new drugs to reduced this risk.

Endothelin is a chemical produced by blood vessels that contributes to the development of hypertension and cardiovascular disease Higher than normal levels of endothelin are seen in patients with vasculitis but how this contributes to cardiovascular disease in patients with vasculitis is not clear. By using drugs that block the effects of endothelin ('endothelin receptor antagonists') the investigators can hopefully reduce the risk of cardiovascular disease in patients with vasculitis. The purpose of the study is to ascertain if endothelin receptor antagonists improve blood vessel function in patients with vasculitis.

DETAILED DESCRIPTION:
Vasculitis patients and healthy controls matched for age, sex will be enrolled into the study. Patients will attend for 4 study days >1 week apart, whereas controls will attend for single day. Circulating Mφ and other immune cells will be confirmed using FACS prior each study.

Study 1 Both patients and control will attend for visit 1: assessment of vascular function using forearm plethysmography as part of case control study.

Vasculitis patients will then attend for visits 2, 3 & 4 as part of randomised three way crossover study (randomised & infusions given in a double-blind method): comparison of the effects of selective ETA receptor antagonism (BQ123; 1000nmol/min for 15min iv), mixed ETA/B antagonism (BQ123/788; 1000 nmol/min & 300 nmol/min for 15 min), and placebo on systemic haemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 years and over
* Body mass index ≤35
* Normal serum albumin

Exclusion Criteria:

* Subject with diabetes or current smoking or chronic kidney disease (eGFR <60ml/min)
* Subject with pre-existing cardiovascular disease
* Subject is below the age of legal consent, or is mentally or legally incapacitated
* History of multiple and/or severe allergic reactions to drugs (including study drugs)
* The subject has donated blood (450 ml) within the last 4 weeks
* Past or present drug or alcohol abuse including intravenous drug abuse at any time
* Participation in another clinical trial within 1 month
* Considered to be at high risk of HIV or hepatitis B
* Women of child-bearing potential (only women who are post-menopausal or surgically-sterilised will be included in the study)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-08; Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Study 1 - forearm blood flow | 20mins
  Response to endothelium-dependent vasodilators
Study 2 - pulse wave velocity | 4 hours
  Response of participants to ET antagonism

SECONDARY OUTCOMES:
Study 1 - tPA release | 20min
  Response of fibrinolytic system to endothelial vasodilators
Study 1 - baseline pulse wave velocity | Baseline
  Baseline arterial stiffness
Study 2 - tPA release | 4 hours
  Response of participants to ET antagonism

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Dhaun, Principal Investigator — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - University of Edinburgh, Edinburgh, Midlothian
  - University of Edinburgh, Edinburgh

REFERENCES:
- [Derived] Farrah TE, Melville V, Czopek A, Fok H, Bruce L, Mills NL, Bailey MA, Webb DJ, Dear JW, Dhaun N. Arterial stiffness, endothelial dysfunction and impaired fibrinolysis are pathogenic mechanisms contributing to cardiovascular risk in ANCA-associated vasculitis. Kidney Int. 2022 Nov;102(5):1115-1126. doi: 10.1016/j.kint.2022.07.026. Epub 2022 Aug 20. PMID 35998848